CLINICAL TRIAL: NCT06507254
Title: MAEVE: Microbiota Mediated Flavonoid Metabolites for Cognitive Health
Brief Title: Polyphenols and Cognitive Decline
Acronym: MAEVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Arpana Church, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB 24-000113; 1R01AG081768 (NIH)
Record Dates: First submitted 2024-05-15; First posted 2024-07-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Decline; Cognitive Dysfunction
Keywords: Polyphenols; Mediterranean Diet; Gut Microbiome; Alzheimers Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyphenol Supplement (Experimental): Juice Plus Essentials, Berry Blend Capsules
  Interventions: Dietary Supplement: Polyphenol Supplement
- Placebo Supplement (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: Polyphenol Supplement — Dietary supplement taken twice daily for 12 months.
  Other Names: Juice Plus Essentials, Berry Blend Capsules
  Arms: Polyphenol Supplement
Dietary Supplement: Placebo Supplement — Dietary supplement taken twice daily for 12 months.
  Arms: Placebo Supplement

SUMMARY:
Globally, populations are aging thereby increasing healthcare burden, overall cognitive impairment, and dementia including Alzheimers diseases (AD). The lack of effective treatments makes it essential to develop new strategies for healthy cognitive aging, including interventions to slow or prevent cognitive decline. A traditional Mediterranean diet, rich in polyphenols (PPs), may prevent or delay the onset of cognitive dysfunction in older adults, preserving healthy brain structure and function, and lowering the risk of AD. These effects, mediated in part by gut microbiome-derived PP metabolites, highlight the role alterations in the brain-gut microbiome system play in neurodegeneration. Moreover, high levels of circulating phenyl-y-valerolactones, neuroprotective compounds, exclusively produced by gut microbiota from flavan-3-ol-rich foods (e.g., cocoa, tea, berries) are associated with delaying the onset of cognitive dysfunction in older adults. Intake of such PPs can also change gut microbial composition and function, altering the physiology of the hosts secondary bile acid (BA) pool, affecting regulatory and signaling functions in the brain as well as cognitive decline and AD. The investigators hypothesize that, in older adults with enhanced AD risk, dietary intake of PPs maintains healthier brain features and cognitive function, and that this beneficial effect is mediated by gut microbiota metabolites of PPs and BAs.

In this multi-PI application by leaders in the field of brain-gut microbiome interactions, the investigators will conduct a year-long, multi-center, randomized double-blind placebo-controlled study in 300 older adults in the United States (validation sample of 100 from Northern Ireland) who are at enhanced risk of developing AD. Ultimately, the investigators will establish the protective effects of regular dietary PP intake on cognitive function and on brain-gut microbiome interactions, ideally allowing the development of effective dietary regimes to prevent of delay the onset of AD in at-risk elderly, thereby reducing cognitive decline and healthcare costs.

Participants will be asked to provide information about their diet, mood, and behaviors via food diaries, physical body measures (e.g. height, weight, etc.), and online questionnaires collected before each in-clinic appointment, as well as monthly online questionnaires. MR imaging will be collected on participants to assess neurocognitive changes as a result of the supplement. Participants will be asked to provide both stool and blood samples. Participants will be randomly assigned to either the Juice Plus+ intervention group or the placebo treatment group and then asked to take their respective supplement 4 pills twice a day. All participants will be asked to come in for 4 in-clinic appointments, including 3 brain MRI scans and 3 cognitive testing appointments, collect 3 stool samples with corresponding diet diaries, and provide 3 blood samples over the course of 12 months. Participants will also meet with a nutritionist 3 times over the 12 months to discuss diet to ensure study eligibility and any questions about the supplement.

ELIGIBILITY:
Inclusion Criteria:

* 50+ Years of age
* Male or Female
* At enhanced risk of Alzheimers Disease (defined as family history of AD, 1st degree family member)
* Overweight or Obese (BMI≥25kg/m^2)
* Habitually consume suboptimal diets such as typical Western Diet (i.e., high in animal products, refined carbohydrates and processed food)
* Able to communicate well in English

Exclusion Criteria:

* Vegan or Vegetarian
* Presence of cognitive impairment at the time of recruitment into the study as measured by the Mini Mental Status Exam (MMSE, score 25-30) and Clinical Dementia Rating (CDR, score=0).
* Pre-existing psychosis or psychiatric conditions
* Currently receiving treatment for dementia
* History of alcohol and/or substance abuse/dependence as determined by a positive endorsement on the MINI+/ If the MINI+ is positive for alcohol or drug dependence, or abuse, the participants will be excluded.
* Heavy use of tobacco (greater than 1/2 pack per day)
* History of cerebrovascular events
* Existing allergies to berry fruits
* Use of oral/IV antibiotics in the last 3 months. Use of probiotics in the last 1 month.
* Recent Changes (last 3 months) in the use of psychoactive medications or other medications that interfere with the measured outcomes.
* Frailty, malnutrition, or food allergy/intolerance requiring special diets.
* Body weight at enrollment greater than 400lbs due to weight restrictions on the MRI table.
* Women who are pregnant, lactating, or postpartum for less than 6months.
* Women of childbearing age who are not practicing birth control or are planning to get pregnant during the study.

Unable to safely participate in the MRI (claustrophobia, presence of devices affected by MRI such as pacemakers, neurostimulators, metallic foreign body, etc.)

* Chronic Pain

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in Polyphenol-derived metabolite concentrations pre, mid, & post intervention - stool | Collected three times by the participant at home, once at baseline (week 0), once at mid-study (month 6), and once at the final 12month appointment (month 12).
  Measurement of metabolomics via stool specimen.
Differences in Polyphenol-derived metabolite concentrations pre, mid, & post intervention - blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Measurement of metabolomics via blood specimen.
Differences in microbiome levels pre, mid, & post intervention - Stool | Collected three times by the participant at home, once at baseline (week 0), once at mid-study (month 6), and once at the final 12month appointment (month 12).
  16S RNA sequencing to measure microbiome levels via stool specimen.
Differences in microbiome levels pre & post intervention - Blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  16S RNA sequencing to measure microbiome levels via blood specimen.
Differences in microbiome levels pre, mid, & post intervention - Stool | Collected three times by the participant at home, once at baseline (week 0), once at mid-study (month 6), and once at the final 12month appointment (month 12).
  Shotgun metagenomics, sequencing to measure microbiome levels via stool specimen.
Differences in microbiome levels pre, mid, & post intervention - Blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Shotgun metagenomics, sequencing to measure microbiome levels via blood specimen.
Differences in Cognitive Measures pre, mid, & post intervention - Executive Function | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Administration of a standardized Stroop Neuro-psychological test; participants ability to correctly identify colors when words are printed in conflicting ink colors.
Differences in Cognitive Measures pre, mid, & post intervention - Executive Function | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Administration of a standardized Trails A & B; participants ability to connect dots, in order, as quickly as possible.
Differences in Cognitive Measures pre, mid, & post intervention | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Differences in Cognitive Measures pre, mid, and post intervention - Executive Functioning | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Administration of a standardized arithmetic task; participants ability to complete quick mental math.

SECONDARY OUTCOMES:
Differences in tryptophan-associated metabolite profiles pre, mid, and post intervention - Stool | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Measurement of tryptophan-associate metabolite profiles via stool specimen.
Differences in Bile Acid's (BA's) pre, mid, & post intervention - Stool | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Measurement of BA's via stool specimen.
Differences in Inflammatory markers pre, mid, & post intervention - Blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Measurement of inflammatory markers via blood specimen.
Differences in Alzheimer's Disease (AD) markers pre, mid, & post intervention - Blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Measurement of AD markers via blood specimen.
Anthropometrics - BMI | Measured three times, once at each in-clinic appointment (week 0, month 6, month 12)
  Measurement of height(in) and weight(lbs), used to calculate body mass index (BMI)
Questionnaire Data | Collected 3 times (1) before beginning the dietary supplement, (2) mid-study month 6, (3) end of study month 12.
  Use of validated surveys to assess ingestive behaviors, social isolation, stress, health, physical activity, etc., self-reported by the participant at home.
Monthly Questionnaire Data | Collected once a month for the duration of the study (12months).
  Use of validated surveys to assess anxiety, depression, stress, and diet, self-reported by the participant at home,
Anthropometrics - waist and hip circumference | Measured three times, once at each in-clinic appointment (week 0, month 6, & month 12)
  Measurement of waist and hip circumference (cm)
Systolic and Diastolic Blood Pressure | Measured three times, once at each in-clinic appointment (week 0, month 6, month 12).
  Measurement of the pressure of circulating blood at rest

OTHER OUTCOMES:
Differences in Multimodal Brain Signatures pre, mid, & post intervention | Measured thrice, once at baseline (week 0), mid-study (month 6), and final 12month appointment (month 12) visit.
  Neuroimaging of participants brain via magnetic resonance imaging (MRI) procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Arpana Church, PhD, Principal Investigator — The Regents of the University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States